CLINICAL TRIAL: NCT02956564
Title: Precision Medical Research of Non-immune Fetal Hydrops (NIFH)-From Prenatal Diagnosis to Intrauterine Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ShanghaiFMIH-FMU1
Record Dates: First submitted 2016-11-02; First posted 2016-11-07 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-11

CONDITIONS: Fetal Hydrops
MeSH Terms: conditions — Hydrops Fetalis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- exposure group (Other): subjects in this group are those who accept intrauterine intervention
  Interventions: Procedure: intrauterine intervention
- control group (No Intervention): subjects in this group are those who do not accept intrauterine intervention

INTERVENTIONS:
Procedure: intrauterine intervention — choose different surgeries according to different causes
  Arms: exposure group

SUMMARY:
Based on multi-center clinical research resources, a large-scale prospective cohort study will be conduted to make a more accurate diagnosis and intervention plan of Non-immune fetal hydrops (NIFH), and then establish NIFH accurate treatment strategy which is suitable for China's national conditions.

DETAILED DESCRIPTION:
1. Etiological study of Non-immune fetal hydrops(NIFH):

   1. Etiological study of NIFH in mid-pregnancy period;
   2. Etiological study of NIFH and hygroma colli in first trimester;
   3. Value assessment of technology for exome sequencing in diagnosis of NIFH;
2. The accuracy of NIFH intrauterine intervention and its effect assessment:

   1. Perinatal outcomes of NIFH ;
   2. The effect of intrauterine treatments.

ELIGIBILITY:
Inclusion Criteria:

* Cases corresponding to diagnosis standards
* Willing to accept the regular follow-up

Exclusion Criteria:

* Immune hydrops fetalis
* Multiple pregnancy, except for twin-to-twin transfusion syndrome IV

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Neonatal mortality | 1 year

SECONDARY OUTCOMES:
Success rate for the operation | 1 week

IPD SHARING:
Plan to Share IPD: Undecided